CLINICAL TRIAL: NCT04368546
Title: Effect of Sunitinib Treatment on Tissue Sodium Accumulation in Patients With Renal Cancer: a Pilot Study
Brief Title: Sunitinib Treatment on Tissue Sodium Accumulation (TSS2)
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Heart Institute (Other)
Responsible Party: Principal Investigator, Dr. Lajos Marko, MD, PhD, Charite University, Berlin, Germany
Other Study IDs: ChariteU-ECRC-TSS2; EA1/044/15 (Other: Ethics Committee of the Charité - Universitätsmedizin Berlin)
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Renal Cell Cancer Metastatic; Hypertension; Sodium Imbalance
Keywords: Sunitinib; Tyrosine kinases-inhibitor; Sodium; MRI; Skin
MeSH Terms: conditions — Hypertension | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Metastatic cell carcinoma patients before sunitinib treatment, after 4 week on, after 2 week off and finally again 4 week on medication.
  Interventions: Drug: Sunitinib
- Healthy controls: Age-matched subjects without known disease.

INTERVENTIONS:
Drug: Sunitinib
  Other Names: Diagnostic test: 23Na-MRI
  Groups: Patients

SUMMARY:
Here, it is investigated how sunitinib, a tyrosine kinase-inhibitor targeting vascular endothelial growth factor receptors, might influence sodium homeostasis in the skin and if this is related to a well-described treatment side-effect of sunitinib, hypertension.

DETAILED DESCRIPTION:
Tyrosine kinases-inhibitors targeting vascular endothelial growth factor (VEGF)-receptors (RTKIs) are increasingly used in oncology in several metastatic tumor types. These agents are featured by toxicities including hypertension. According to a new insight, sodium in response to a high dietary sodium intake, is accumulated in a hyperosmolar way in the interstitial compartment. In response to this high sodium concentration cells of the mononuclear phagocytic system (MPS) are activated resulting in an increased production of VEGF-C, activation of VEGF type 3 receptors and formation of a lymphatic capillary network, involved in clearance of interstitial sodium. Blockade of stimulation of VEGF-C receptors or depletion of MPS cells in rodents has been associated with salt-sensitive hypertension.

Sunitinib is an orally-active, multitarget RTKI mainly used for the treatment of patients with metastatic renal cancer and imatinib-resistant gastrointestinal stromal tumors. Sunitinib blocks all three VEGF receptors subtypes, including VEGF-receptor type 3.

The investigators hypothesize that treatment of patients with sunitinib is associated with tissue sodium accumulation and this accumulation contributes to the rise in blood pressure. Tissue sodium is measured by using a newly developed 23Na magnetic resonance-imaging (MRI) technique which allows a non-invasive and contrast agent-free sodium content measurement in the muscle and skin of the lower leg.

ELIGIBILITY:
Inclusion Criteria:

* Age men > 18 years
* Life-expectation > 3 months
* Stable weight
* Blood pressure below 140/90 mmHg at baseline
* Estimated glomerular filtration rate > 45 ml/min/1.73m2
* Willingness to give written informed consent

Exclusion Criteria:

* Heart failure
* Liver disease with ascites
* Nephrotic syndrome
* Gastrointestinal complaints, preventing normal daily food intake or diarrhea
* Any form of diabetes mellitus
* Known autoimmune diseases
* Acute or chronic infection
* Alcohol or substance abuse

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The effect of the female hormonal cycle on skin sodium homeostasis is unknown, therefore we include here male subjects only.
Study Population: Patients with metastatic renal cell carcinome in the primary care of the Charité - Universitätsmedizin Berlin as well as healthy subjects without known disease recruited in the Charité - Universitätsmedizin Berlin and healthy volunteers form the Max-Delbrück Center of Molecular Medicine
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Skin sodium | 3 months (before, 4 weeks on, 2 weeks off and 4 weeks on medication)
  Changes in sodium content measured by 23Na magnetic resonance-imaging (MRI) technique

SECONDARY OUTCOMES:
Plasma VEGF-C | 3 months (before, 4 weeks on, 2 weeks off and 4 weeks on medication)
  Concentration of VEGF-C in patients plasma

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Müller, PhD, Study Director — Group leader at the Max Delbruck Center for Molecular Medicine
Locations (1):
- Experimental and Clinical Research Center, Clinical Research Unit, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kandula P, Agarwal R. Proteinuria and hypertension with tyrosine kinase inhibitors. Kidney Int. 2011 Dec;80(12):1271-7. doi: 10.1038/ki.2011.288. Epub 2011 Sep 7. PMID 21900879
- [Background] Kappers MH, van Esch JH, Sluiter W, Sleijfer S, Danser AH, van den Meiracker AH. Hypertension induced by the tyrosine kinase inhibitor sunitinib is associated with increased circulating endothelin-1 levels. Hypertension. 2010 Oct;56(4):675-81. doi: 10.1161/HYPERTENSIONAHA.109.149690. Epub 2010 Aug 23. PMID 20733093
- [Background] Machnik A, Neuhofer W, Jantsch J, Dahlmann A, Tammela T, Machura K, Park JK, Beck FX, Muller DN, Derer W, Goss J, Ziomber A, Dietsch P, Wagner H, van Rooijen N, Kurtz A, Hilgers KF, Alitalo K, Eckardt KU, Luft FC, Kerjaschki D, Titze J. Macrophages regulate salt-dependent volume and blood pressure by a vascular endothelial growth factor-C-dependent buffering mechanism. Nat Med. 2009 May;15(5):545-52. doi: 10.1038/nm.1960. Epub 2009 May 3. PMID 19412173
- [Background] Kopp C, Linz P, Dahlmann A, Hammon M, Jantsch J, Muller DN, Schmieder RE, Cavallaro A, Eckardt KU, Uder M, Luft FC, Titze J. 23Na magnetic resonance imaging-determined tissue sodium in healthy subjects and hypertensive patients. Hypertension. 2013 Mar;61(3):635-40. doi: 10.1161/HYPERTENSIONAHA.111.00566. Epub 2013 Jan 21. PMID 23339169